CLINICAL TRIAL: NCT06275841
Title: A PHASE 1, OPEN-LABEL, 2-PERIOD STUDY TO EVALUATE THE EFFECT OF MULTIPLE DOSES OF ESOMEPRAZOLE ON THE PHARMACOKINETICS OF SINGLE DOSE VEPDEGESTRANT (ARV-471, PF-07850327) UNDER THE FED CONDITION IN HEALTHY ADULT MALES AND HEALTHY ADULT FEMALES OF NONCHILDBEARING POTENTIAL
Brief Title: A Study to Learn If the Study Medicine Esomeprazole Changes How the Body Processes the Other Study Medicine Vepdegestrant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4891035
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- vepdegestrant with or without esomeprazole (Experimental): vepdegestrant administered as a single dose in Period 1 and Period 2. Esomeprazole administered once a day for 5 days in Period 2
  Interventions: Drug: vepdegestrant; Drug: esomeprazole

INTERVENTIONS:
Drug: vepdegestrant — experimental
Drug: esomeprazole — Experimental treatment to assess an endpoint

SUMMARY:
The purpose of the study is to investigate the effect of multiple doses of a proton-pump inhibitor (PPI) esomeprazole on the PK of vepdegestrant under fed conditions in healthy adult participants.

All participants in this study will receive one dose of vepdegestrant alone by mouth in Period 1. In Period 2, everyone will receive esomeprazole by mouth once a day for multiple days. Participants will also receive one dose of vepdegestrant by mouth. The levels of vepdegestrant in Period 1 will be compared to the levels of vepdegestrant in Period 2 to determine if the PPI affects how vepdegestrant is processed differently in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male participants, and female participants of non-childbearing potential, aged 18 years or older (or the minimum age of consent in accordance with local regulations) at Screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs and standard 12-lead ECGs.
* BMI of 16-32 kg/m2; and a total body weight >45 kg (99.2 lb).
* Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in the ICD and in this protocol.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Breastfeeding female participants; Male participants with partners currently pregnant; fertile male participants who have partners of childbearing potential and are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for 30 days after the last dose of investigational product.
* Participants with known history of sensitivity to vepdegestrant or esomeprazole or any of the formulation components of vepdegestrant or esomeprazole.
* Use of prescription or nonprescription drugs and/or dietary and/or herbal supplements and/or vitamins within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention. (Refer to Section 6.9 Prior and Concomitant Therapy for additional details). A longer washout is required for those that fall into the categories below:

  * Acid-reducing agents such as PPI (except as study drug administered) must be discontinued at least 14 days prior to the first dose of study intervention.
  * Moderate or strong CYP3A inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
  * Moderate or strong CYP3A inhibitor which are prohibited within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test. A single repeat for positive drug screen may be allowed.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm/Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Renal impairment as defined by an eGFR <60 mL/min/1.73 m2. Based upon participant age at Screening, eGFR is calculated using the recommended formulas in Section 10.7.2 to determine eligibility and to provide a baseline to quantify any subsequent kidney safety events.

For eligibility assessment based upon estimated renal function, the higher of the Screening and baseline eGFR values may be used.

* Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If QTcF exceeds 450 ms, or QRS exceeds 120 ms, the ECG should be repeated twice and the average of the 3 QTcF or QRS values used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
* Participants with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  • ALT, AST, or Total Bilirubin Level ≥1.5 × ULN.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
* History of use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of vepdegestrant when vepdegestrant is administered alone | Period 1 - Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Maxium observed plasma concentration of vepdegestrant when vepdegestrant is administered with esomeprazole | Period 2 - Day 5 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Area under the curve from time zero to extrapolated infinite time (AUCinf) when vepdegestrant is administered alone | Period 1 - Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
  AUCinf=area under the plasama concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time. It is obtained from AUC (0-t) plus AUC (t-inf)
Area under the curve from time zero to extrapolated infinite time (AUCinf) when vepdegestrant is administered with esomeprazole | Period 2 - Day 5 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
  AUCinf=area under the plasama concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time. It is obtained from AUC (0-t) plus AUC (t-inf)

SECONDARY OUTCOMES:
number of participants with treatment-emergent adverse events (AEs) and serious adverse events (SAEs) | time the participant provides informed censent through and including follow-up contact occurring 28-35 calendar days after the last administration of the study intervention
  An AE is any untoward medical occurence in a participant who received study drug without regard to possibility of causal relationship with the study treatmnet. SAE is defined as one of hte following: is fatal or life-threatening; results in persistent or significant disability/incapacity; constitues a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE is defined as an AE with onset data occurring during the on-treatment period. AEs include all SAEs and non-SAEs.
Number of participants with clinical laboratory abnormalities | baseline up to Period 2 Day 12
  Following parameters were analyezed for laboratory examination: hematology (Hemoglobin, Hematocrit, RBC count, Platelet count, WBC count, Total neutrophils, Eosinophils, Monocytes, Basophils, Lymphocytes); liver function (AST, ALT, Total bilirubin, Alkaline phosphatase, Albumin, Total protein); renal function (blood Urea nitrogen, Creatinine, Cystatin Ca, uric acid); eletrolytes (Calcium, Sodium, Potassium Chloride, Total CO2 (bicarbonate)); clinical chemistry (glucose); urinalysis (dipstick [decimal logarithm of reciprocal of hydrogen ion activity [pH] of urine, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, bilirubin], microscopy
  If Hb/RBC abnormal:
  MCV, MCH, MCHC
  )
Number of participants with electrocardiogram (ECG) abnormalities | Baseline up to Period 2 Day 12
  ECG abnormalities criteria include 2) a postdose QTcF is increased by >60 ms from the baseline and is >450 ms; or b) an absolute QTcF value is >500 ms for any scheduled ECG.
Number of participans with clinically significant change from baseline in vital signs | Baseline up to Period 2 Day 12
  Blood pressure and pulse rate will be performed following at least a 5-minute rest in a supine position

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891035